CLINICAL TRIAL: NCT06836115
Title: Reading Problems and Stuttering
Brief Title: Reading and Stuttering
Status: Not yet recruiting | Type: Observational
Sponsor: Wafaa Helmy Abdelhakeem (Other)
Responsible Party: Sponsor-Investigator, Wafaa Helmy Abdelhakeem, doctor, Minia University
Organization: Minia University (Other)
Other Study IDs: reading problems in stuttering
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group A: will include with 100 participants with developmental stuttering
- group B: will include 100 participants with normal fluency speech.

SUMMARY:
Dyslexia is a common neurodevelopmental condition, which manifests itself in the form of reading difficulties and occurs in 7-10% of the population (Peterson & Pennington, 2012).

As for dyslexia, it is one of the most common learning disorders and the most common cause of difficulties with reading, writing, and spelling. The global prevalence of dyslexia is estimated to be between 5% and 10% of the population, but it may be as high as 17% (Sprenger-Charolles et al., 2011). Stuttering is a speech disorder characterized by involuntary, audible, or silent repetitions or prolongations of sounds or syllables, along with disturbances in the fluency of verbal phrases.Stuttering and dyslexia are two processing deficits that have an impact on a person's social and academic lives, especially as they usually affect the pediatric population more than adults. Even though they affect different domains, they have similar characteristics in their pathogenesis, epidemiology, and impact on life (Algaidy et al., 2023). The aim of the study will be to identify the prevelance of dyslexia in developmental stuttering.

ELIGIBILITY:
Inclusion Criteria:

* children with stuttering

Exclusion Criteria:

* children with delayed language development

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will include 200 patients. Subjects will be divided into two groups, group A will include with 100 participants with developmental stuttering and group B will include 100 participants with normal fluency speech.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
4- Arabic Reading Test | baseline
  arabic reading test in scores

IPD SHARING:
Plan to Share IPD: Undecided